CLINICAL TRIAL: NCT06823661
Title: Feasibility and Acceptability of Transcutaneous Electrical Stimulation for Apnea Detected by Capnography (TESCapno): A Pilot Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Stimulation for Apnea Detected by Capnography
Acronym: TESCapno
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Mohammad Goudarzi Rad, RN, PhD Candidate, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 55095
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Depression; Opioids
Keywords: respiratory depression; Capnography; sedation; Transcutaneous electrical nerve stimulation (TENS)
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients, PACU nurses, and other healthcare providers (anesthesiologists and surgeons) will be kept unaware of the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Electrical Stimulation (TES) (Experimental): All patients assigned to the intervention group will be continuously monitored by capnography, which is attached to the TES device. This monitoring will continuously track end-tidal carbon dioxide (ETCO2) levels. A mild electrical stimulation will be initiated when the episode of apnea ≥10 seconds is detected by the capnography. Patients in the intervention group will receive TES applied to the ventral surface of the forearm via electrodes in response to the apnea lasting for more than or equal to 10 seconds. When apnea persists for more than or equal 10 seconds, a pre-determined, patient-specific mA current stimulus will be administered for one second. If the patient has not taken a breath after the first stimulation, a second stimulus of similar intensity will be administered for three seconds. Subsequently, all stimuli will be administered for three seconds until the apnea criteria have ceased.
  Interventions: Device: transcutaneous electrical nerve stimulation (TENS)
- Placebo (Monitor-Only mode) (No Intervention): The control group will be monitored by capnography attached to the TES device. The TES electrode will be placed on the ventral surface of the wrist, but no stimulus will be applied (Monitor-Only mode). Participants in the control group will be checked during the PACU stay to make sure that they are still comfortable, and any adverse events will be documented.

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation (TENS) — A TENS 3000-unit, which is FDA and health Canada approved (Licence No.: 95655) and operated by a small 9V block battery will be used. Potential participants will receive a detailed written explanation of the TES protocol and a brief demonstration of how it works, including the feeling produced by the skin stimulator. Patient-specific TES thresholds will be determined after informed written consent for study participation is obtained. Surface electrode pads will be placed on the ventral surface of the forearm, and 1-Hz pulses will be gradually administered with an increase in current. Patients will be asked to report when they first feel the stimulation and when it becomes annoying. The milliamp current associated with these two levels of stimulation will be recorded on the participant's baseline data collection form. The "annoying" thresholds for all study participants will be used to deliver stimuli in response to respiratory depression in the PACU.
  Arms: Transcutaneous Electrical Stimulation (TES)

SUMMARY:
After surgery, patients often recover in a special area called the Post Anesthesia Care Unit (PACU). Patients may receive pain medications either during the surgery or afterward in the PACU. While these medications are important for controlling pain, some of them can slow down breathing.

To ensure patients' breathing remains safe, the nurses in the PACU monitor respiratory rate (how many breaths a patient takes per minute) and oxygen levels using standard monitoring equipment. This is the usual way they check for breathing concerns. If these monitors show that a patient's breathing has slowed down too much, nurses may wake the patient up or stimulate them using their voice or gentle physical touch to encourage deeper breaths.

What is this study about? This research is testing a new approach that uses an additional monitor called capnography. Capnography helps detect slowing or stopping of breathing by measuring the carbon dioxide (CO2) exhaled by patients. If the monitor shows slowed or stopped breathing (called apnea, lasting at least 10 seconds), this study will test using a technology called transcutaneous electrical stimulation (TES) to encourage normal breathing.

How does TES work? TES provides a slight, annoying sensation on the patient's skin-enough to wake them up without causing pain. This has been used in other studies to safely restore breathing after surgery. In this study, the researchers are testing whether a new automated device can deliver TES when the capnography monitor detects breathing issues. The goal is to test the feasibility (can this system work in the PACU?) and acceptability (how do patients feel about this approach?) of this technology.

Who can join this study? Adults aged 18 or older who received general anesthesia and medications (opioids) for pain control during or after surgery are eligible. Patients recovering from surgery in the PACU at Toronto General Hospital may be invited to participate.

Why is this study important? The study aims to reduce the risk of opioid-related breathing problems after surgery, making recovery safer and more comfortable for patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years old
* Adults undergoing an elective (General, Plastics, Urology, Gynecologic Oncology, Vascular, Otolaryngology, Transplant) surgery with general anesthesia who are recovering in the PACU
* American Society of Anesthesiologists (ASA) grade I-IV
* Scheduled to be seen at the Pre-Admission Clinic or Surgery Inpatient Unit
* Able to complete questionnaires with or without assistance
* Able to understand the study protocol, its requirements, risks, and discomforts
* Able to provide written informed consent

Exclusion Criteria:

* A) Preoperative exclusion criteria:

  * American Society of Anesthesiologists (ASA) grade V-VI
  * Urgent or emergent surgical procedures that there is insufficient time prior to anticipated commencement of the procedure for participation in the study
  * Patients with implantable medical electronic devices (eg, pacemaker, implantable cardioverter defibrillator, catheter, and so on.)
  * Patients with febrile illnesses or acute infectious diseases
  * Pregnancy
  * Epilepsy.
* B) Postoperative exclusion criteria:

  * Surgery that would preclude the use of a nasal cannula or face mask used for capnography monitoring (e.g., facial reconstruction)
  * Postoperative mental status precludes application of study equipment, including a nasal cannula/face mask and/or the stimulation pads (e.g., delirium or agitation during recovering from anesthesia, repeated removal of cannula)
  * Postoperative admission to the ICU or any site other than the PACU
  * Need for postoperative assisted ventilation via an endotracheal tube or tracheostomy
  * An abnormal respiratory tract identified during or immediately after surgery can lead to severe respiratory obstruction
  * Patients with cardiac arrhythmia (history of atrial fibrillation or bundle branch block)
  * Skin conditions such as open sores preventing proper application of electrodes
  * Presence of metal implants in both arms
  * Lack of access to upper extremities following surgery for application of the stimulation pads

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Up to an hour after PACU admission
  Recruitment in the TES pilot trial is defined as the number of eligible study participants who agreed to participate in this pilot trial compared to the total number of eligible participants who met the inclusion criteria. The Participant Recruitment and Follow-Up Form will be completed by the researcher and used to track recruitment procedures (i.e., recruitment rates and reasons for participation and non-participation). Participants are not required to provide a reason for declining to participate in the research. However, if they choose to share their reasons, we will note their reasons for refusal.
Retention | Up to an hour after PACU admission
  Retention is defined as the number of participants who enroll and stay in this pilot trial through completing the follow-up assessment at the end of the observation period among the total trial participants. This variable is measured using the Participant Recruitment and Follow-Up Form. The form has the following items: TESCapno trial ID, completing pain assessment, TES and opioid related adverse events form in both groups.
Acceptability | Up to an hour after PACU admission
  Acceptability of the intervention will be assessed using the Intervention Acceptability Form and will be completed by participants at the end of observation period. Acceptability of the TES is a self-report questionnaire developed by the researchers containing 5-point Likert scales: 1= "strongly disagree"; 2= "disagree"; 3= "neutral"; 4= "agree"; 5= "strongly agree". Responses to Likert scale questions will be reported using means and standard deviations. In the absence of reference interpretations of the acceptability questionnaire, the midpoint of Likert scale will be selected as the minimum level of acceptability of the TES device.

SECONDARY OUTCOMES:
1. Duration of 'apnea' | Up to an hour after PACU admission
  Apnea is defined as the cessation of breathing for a minimum of 10 seconds, and it's the most repetitive feature of opioid-induced respiratory depression (OIRD) in postoperative patients. Therefore, for the purpose of this study, the cumulative duration of detected apnea events lasting ≥ 10 seconds over the duration of recording in both groups will be captured using continuous capnography measurements with the Capnostream device. The Capnostream™ 20p monitor (Medtronic) will be used to offer "real-time" observation of apnea.
2. Incidence of respiratory depression | Up to an hour after PACU admission
  During the observation period, the incidence of RD episodes in the PACU will be captured by continuous capnography and pulse oximetry measurements and recorded to a laptop in conjunction with the clinical data as reported by the research student. The clinical data and monitor parameters specified below are considered an episode of RD:
  * EtCO2 ≤ 15 or ≥ 60 mmHg for ≥ 3 minutes.
  * RR ≤ 5 breaths for ≥ 3 minutes.
  * SpO2 ≤ 85% for ≥ 3 minutes.
  * Apnea episode lasting ≥ 30 seconds
  * Any respiratory opioid-related adverse drug event (rORADE)
3. Nursing interventions to manage respiratory depression | Up to an hour after PACU admission
  During the observation period, nursing interventions aimed at addressing respiratory depression include providing verbal instructions to encourage breathing, physically stimulating the patient, employing a stir-up regimen (repositioning, coughing, deep breathing, and incentive spirometry), and increasing or adding supplemental oxygen will be recorded.
  A researcher-designed questionnaire will be used to evaluate the nursing interventions aimed at addressing respiratory depression. This questionnaire will assess the implementation of interventions, such as verbal stimulation, tactile stimulation, the stir-up regimen (repositioning, coughing, deep breathing, and incentive spirometry), and the use of increased or supplemental oxygen.
4. TES-related adverse events | Up to an hour after PACU admission
  At the end of the observation period, the researcher will inspect participants' skin integrity around the TES region to assess for anticipated and unanticipated adverse events in the all groups. The adverse events will be considered as painful sensations or other uncomfortable reactions, including cutaneous injuries, unresolved numbness, tingling of extremity, skin irritation, tenderness or soreness, and discomfort.
5. Pain level | Up to an hour after PACU admission
  Before starting the intervention and at the end of the observation period, subjective pain assessments will be performed using a visual analog scale (VAS). The VAS utilizes a 100-mm horizontal line, marked from 0 to 10 from left to right, where zero represents 'no pain' and 10 represents the 'worst possible pain.' Participants will be asked by the researcher to indicate on the line the point that corresponds to their perception of their current pain level. This scale allows for the measurement of pain, which can range across a continuum from no pain to the most severe pain imaginable. The VAS is easy to use, valid and reliable compared with other pain rating scales (r=.71-.78, intraclass correlation coefficient [ICC]=.71-.99).
6. Total opioids consumption | Up to an hour after PACU admission
  At the end of observation period, intraoperative and postoperative administration of opioids will be recorded and then converted to total morphine milligram equivalents (MME), a standardized unit that allows for comparison across different opioid types. This is done by multiplying the quantity and dose, and applying standard conversion tables.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto

IPD SHARING:
Plan to Share IPD: No
All study data will be managed in accordance with the Tri-Agency principles of health data management and according to P-HIPPA guidelines. No personal identifiable information will be collected. The electronic demographic questionnaires will contain no personal identifiers and will also be stored on an encrypted UHN laptop. The master participants list is a document that maintains a confidential list of names of all subjects participating in the clinical study. It links each patient to a unique ID number to be used on all data forms in the study. To access all the electronic files, there will be a password to login to the laptop and a different password to access the UHN OneDrive. Study-related documents (e.g., signed informed Participant Information and Consent Form (PICF)) data will be locked and only the study team will have access. All raw data collected at Toronto General Hospital - University Health Network will be stored at the organization at the end of the study.

REFERENCES:
- [Background] Khanna AK, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Lee S, Ti LK, Urman RD, McIntyre R Jr, Tornero C, Dahan A, Saager L, Weingarten TN, Wittmann M, Auckley D, Brazzi L, Le Guen M, Soto R, Schramm F, Ayad S, Kaw R, Di Stefano P, Sessler DI, Uribe A, Moll V, Dempsey SJ, Buhre W, Overdyk FJ; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Collaborators. Prediction of Opioid-Induced Respiratory Depression on Inpatient Wards Using Continuous Capnography and Oximetry: An International Prospective, Observational Trial. Anesth Analg. 2020 Oct;131(4):1012-1024. doi: 10.1213/ANE.0000000000004788. PMID 32925318
- [Background] DeLoach LJ, Higgins MS, Caplan AB, Stiff JL. The visual analog scale in the immediate postoperative period: intrasubject variability and correlation with a numeric scale. Anesth Analg. 1998 Jan;86(1):102-6. doi: 10.1097/00000539-199801000-00020. PMID 9428860
- [Background] Dahan A, van der Schrier R, Smith T, Aarts L, van Velzen M, Niesters M. Averting Opioid-induced Respiratory Depression without Affecting Analgesia. Anesthesiology. 2018 May;128(5):1027-1037. doi: 10.1097/ALN.0000000000002184. PMID 29553984
- [Background] ELECTROPHYSICAL AGENTS - Contraindications And Precautions: An Evidence-Based Approach To Clinical Decision Making In Physical Therapy. Physiother Can. 2010 Fall;62(5):1-80. doi: 10.3138/ptc.62.5. Epub 2011 Jan 5. No abstract available. PMID 21886384